CLINICAL TRIAL: NCT02327806
Title: The Effect of Pullsed Magnetic Field Induction on Improving the Forearm Tissue Muscle Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 483-14-TLV
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Medical Oncology

ARMS (3):
- 10 minutes of pulsed electromagnetic field therapy (Other): 10 minutes of pulsed electromagnetic field therapy
  Interventions: Device: pulsed electromagnetic field therapy
- 20 minutes of pulsed electromagnetic field therapy (Other): 20 minutes of pulsed electromagnetic field therapy
  Interventions: Device: pulsed electromagnetic field therapy
- 30 minutes of pulsed electromagnetic field therapy (Other): 30 minutes of pulsed electromagnetic field therapy
  Interventions: Device: pulsed electromagnetic field therapy

INTERVENTIONS:
Device: pulsed electromagnetic field therapy

SUMMARY:
Pulsed electromagnetic field therapy (PEMFT) is a reparative technique most commonly used in the field of orthopedics for the treatment of non-union fractures. The aim is to test the effect of the magnetic induction on brute force of treated muscle in oncological patients. Oncology patients were chosen as we assume that the ipmrovement will be more noticable in oncology patients than in a non-oncology, healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patiant from the oncology clinic

Exclusion Criteria:

* Known bone disease
* Pregnancy
* Birth defects or acquired uper extremity
* Neurology disease
* Medical history in the forehand
* Pacemaker neural modulation pacer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Brute force | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Unit, Sourasky Medical Center, Tel Aviv, Israel